CLINICAL TRIAL: NCT02379026
Title: Improving Body Composition, Strength, Function and Health Related Quality of Life in Older Individuals With Sarcopenic Obesity Through Lifestyle Modifications
Brief Title: Lifestyle Modifications for the Treatment of Sarcopenic Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Margaret University (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Christos Theodorakopoulos, Mr, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QueenMU
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Sarcopenic Obesity; Sarcopenia; Obesity
MeSH Terms: conditions — Sarcopenia; Obesity | interventions — Exercise; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise & Protein Drink/Diet (Experimental): High-protein (1.2-1.5 g protein per kg bodyweight; a milk-based protein drink will provide 50 g protein/day) energy-restricted (500 kcal deficit) diet and a multimodal exercise program (balance, flexibility, aerobic, resistance) 3 times/week, each lasting 1 hour. 1 tablet of Vitamin D3 (25 micrograms) x three days/week. Total duration 16 weeks.
  Interventions: Dietary Supplement: Protein Drink/Diet; Behavioral: Exercise; Dietary Supplement: Vitamin D3
- Exercise (Active Comparator): A multimodal exercise program (balance, flexibility, aerobic, resistance) will take place 3 times/week, each one lasting 1 hour. Participants in this group will follow their habitual diet. 1 tablet of Vitamin D3 (25 micrograms) x three days/week. Total duration 16 weeks.
  Interventions: Behavioral: Exercise; Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Protein Drink/Diet — 1.2 - 1.5 g of protein per kilogram bodyweight will be consumed per day. One milk-based beverage high in dairy protein (50g of protein per 500ml bottle) will be consumed every day (post-workout on exercise days, before bed on non-exercise days). A 500kcal deficit diet will be prescribed based on the individual characteristics (eg weight, age, physical activity levels) of each participant.
  Arms: Exercise & Protein Drink/Diet
Behavioral: Exercise — Participants will enrol in a multimodal exercise program (with balance, flexibility, resistance and aerobic elements) 3 times a week, each lasting 1 hour.
Dietary Supplement: Vitamin D3 — 1 tablet of Vitamin D3 (25 micrograms) will be taken on 3 non-consecutive days/ week to achieve a weekly intake of 75 micrograms.

SUMMARY:
This study evaluates the addition of a high-protein energy-restricted diet to exercise in the treatment of sarcopenic obesity in people aged 65 and over. Half of participants will follow a hypocaloric (500 kcal deficit) high-protein (1.2 -1.5 g Protein/ kg bodyweight) diet alongside an exercise regime, while the other half will follow the same exercise regime alongside their habitual diet . All participants will consume a Vitamin D3 tablet (25micrograms) 3 times a week to achieve a weekly intake of 75 micrograms. Total duration of the intervention will be 16 weeks.

DETAILED DESCRIPTION:
Sarcopenic Obesity is associated with advanced ageing and is characterised by increased adipose tissue and loss of muscle mass, strength and/or function. The combination of sarcopenia and obesity can predispose older individuals to more functional disabilities than either of these two conditions alone, leading eventually to increased rates of morbidity and mortality. Lifestyle interventions focusing on physical activity and diet have been suggested as an effective tackling strategy. However, there is limited evidence on the efficacy of such interventions in sarcopenic obese individuals over 65 years of age. Therefore, the aim of this study is to assess the impact of a high protein energy-restriction diet and a mixed exercise program on body composition, strength, functionality and quality of life in older people with sarcopenic obesity.

This is a prospective randomised control trial among independent living sarcopenic obese community-dwellers. Eligible participants are people over 65y who experience increased adiposity (% body fat >28% in men and >40% in women) and low skeletal muscle index (SMI <10.75 kg/m2 in men and <6.75kg/m2 in women). Fifty (50) participants will be randomly allocated to either the exercise group (EX) or the exercise plus high protein energy-restricted diet group (EXD). Each group will undergo 3 exercise sessions/ week for a period of 16 weeks. The exercise sessions will be similar for both groups and will incorporate aerobic, resistance, balance and flexibility elements. The EXD group will receive a 500kcal-deficit diet plan and a milk-based protein supplement (ProMilk 50 by Myprotein; 50 g milk protein/ 500 ml bottle) to consume every day (at post-workout on exercise days or as a pre-bed snack on non-exercising days). The protein consumption will be in the range of 1.2-1.5 g.kg bw-1. A total weekly dose of 75mcg Vitamin D3 (3 x 25mcg) will be administered orally to all participants to avoid potential confounders associated with Vitamin D deficiency/hypovitaminosis. The primary and secondary outcomes will be evaluated at baseline, week 10 and week 16.

ELIGIBILITY:
Inclusion Criteria:

* Independent living community-dwellers
* Sarcopenic
* Obese
* Montreal Cognitive Assessment test (MoCA) score > or = 26

Exclusion Criteria:

* Use of pacemaker
* Lactose intolerance
* Parkinson's disease
* Unmanaged pain
* Severe osteoporosis or arthritis
* Use of corticosteroids
* History of pulmonary embolus or myocardial infarction within the previous 2 years
* Heart disease
* Chronic obstructive pulmonary disease
* Chronic kidney disease
* Hypertension (resting systolic pressure >200mmHg, resting diastolic >100mmHg)
* Acute systemic illnesses
* Any other uncontrolled physical, psychological or mental condition that either prohibits adherence to the study protocol or increases significantly the health risks for the subject.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle mass | Baseline, 10 weeks, 16 weeks
  Assess changes in total skeletal muscle mass (in kilograms) using bioelectrical impedance analysis at baseline, week 10 and week 16.
Body fat mass | Baseline, 10 weeks, 16 weeks
  Assess changes in body fat mass (in kg) using bioelectrical impedance analysis at baseline, week 10 and week 16.

SECONDARY OUTCOMES:
Physical Performance | Baseline, 10 weeks, 16 weeks
  Assess changes in Physical performance using the Short Physical Performance Battery test (SPPB) with a maximum score of 12.
Dynamic Balance | Baseline, 10 weeks, 16 weeks
  Assess changes in dynamic balance using the 1-Arm Reach test (measured in cm).
Functional Mobility | Baseline, 10 weeks, 16 weeks
  Assess changes in functional mobility using the timed (in seconds) Get Up-and-go test for 6 meters.
Health related quality of life | Baseline, 16 weeks
  Assess changes in health related quality of life using the Rand SF-36 questionnaire.
Central adiposity | Baseline, 10 weeks, 16 weeks
  Assess changes in central adiposity by measuring the Sagittal Abdominal Diameter (in cm)
Handgrip strength | Baseline, 10 weeks, 16 weeks
  Assess changes in handgrip strength (in kg) using a handgrip dynamometer

OTHER OUTCOMES:
Dietary intake | Baseline, 16 weeks
  Assess changes in dietary intakes using 3-day recorded diet diaries from baseline to week 16
Serum vitamin D (25-OH) levels | Baseline, 16 weeks
  Assess changes in serum vitamin D levels at baseline and week 16

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Bannerman, PhD, Study Director — Queen Margaret University
Locations (1):
- Queen Margaret University, Musselburgh, United Kingdom